CLINICAL TRIAL: NCT03371108
Title: AN OPEN-LABEL, RANDOMIZED, MULTICENTER, PHASE 3 STUDY TO COMPARE THE IMMUNOGENICITY, EFFICACY, AND SAFETY OF GAN & LEE PHARMACEUTICALS INSULIN GLARGINE INJECTION TO LANTUS® IN ADULT SUBJECTS WITH TYPE 2 DIABETES MELLITUS
Brief Title: Gan & Lee Insulin Glargine Target Type (2) Evaluating Research
Acronym: GLITTER 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GLAT2-3002
Record Dates: First submitted 2017-11-20; First posted 2017-12-13 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Diabetes Type 2; Type 2; Basal; Insulin; Glargine; T2DM; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — gallium nitrate; Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Subjects who meet the study eligibility criteria will be centrally randomized 1:1 in an open-label fashion to receive either Gan & Lee Insulin Glargine Injection or Lantus® for 26 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gan & Lee Insulin Glargine Injection (Experimental): Gan & Lee Insulin Glargine Injection solution for subcutaneous injection, 100 U/mL, in the integrated, disposable 3.0 mL prefilled Gan & Lee injector pen. Subjects randomized to the Gan & Lee Insulin Glargine Injection group will participate in the study for 26 weeks.
  Interventions: Biological: Gan & Lee Insulin Glargine Injection
- Lantus® (Active Comparator): Lantus® solution for subcutaneous injection, 100 U/mL, in the SoloStar® 3.0 mL prefilled insulin pen. Subjects randomized to the Lantus® group will participate for 26 weeks.
  Interventions: Biological: Lantus®

INTERVENTIONS:
Biological: Gan & Lee Insulin Glargine Injection — Route of administration: subcutaneous injection
  Arms: Gan & Lee Insulin Glargine Injection
Biological: Lantus® — Route of administration: subcutaneous injection
  Arms: Lantus®

SUMMARY:
Primary Objective:

• To evaluate equivalence of Gan & Lee Insulin Glargine Injection and Lantus® in terms of immunogenicity

Secondary Objective:

Immunogenicity:

• To evaluate the percentage of subjects with negative anti-insulin antibodies (AIA) at baseline who develop confirmed positive AIA up to Week 26, the percentage of subjects with at least a 4-fold increase in titers compared to baseline value, mean change from baseline in AIA titers between treatment groups, the percentage of subjects with confirmed positive AIA who develop any anti-insulin neutralizing antibodies up to visit Week 26, and the percentage of subjects in each treatment group with confirmed positive AIA up to visit Week 26

Safety:

• To evaluate the safety of Gan & Lee Insulin Glargine Injection in comparison with that of Lantus®

Efficacy:

• To evaluate the efficacy of Gan & Lee Insulin Glargine Injection in comparison with that of Lantus®

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant, nonlactating female subjects between the ages of 18 and 75 years, inclusive.
2. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH GCP Guideline E6 and all applicable regulations, before initiating any study related procedures.
3. Ability to understand and fully comply with all study procedures and restrictions.
4. Subjects with a confirmed diagnosis of type 2 diabetes mellitus who meet one of the following:

   1. If insulin-naïve, subjects should have been on at least 2 approved OAMs for at least 12 weeks before screening, and the clinician has decided to add insulin therapy.
   2. If already being treated with a basal and/or bolus insulin, subjects should have been treated with insulin for at least 6 months in addition to at least 1 approved OAM, and must not have changed the type or brand of insulin within 6 months prior to screening.
5. HbA1c values as follows:

   1. If insulin-naïve, HbA1c ≤ 11.0%.
   2. If previously on a basal insulin regimen, HbA1c ≥ 7.0% and ≤ 11.0%.
6. Body mass index (BMI) ≤ 45 kg/m2.
7. Adherence to a prudent diet and exercise regimen recommended by the medical provider, and willingness to maintain these consistently for the duration of the study.
8. Concomitant medications are allowed, provided that no significant dosing changes are anticipated during the study (see the exclusion criteria below for specific prohibited concomitant medications); for concomitant thyroid medications, subjects must have been on a stable dosage for 90 days before screening.

Exclusion Criteria:

1. Participation in another clinical study or use of any study drug within 30 days before screening.
2. Previous use of a biosimilar insulin, either basal or bolus.
3. Diabetic ketoacidosis within a year before screening.
4. Brittle type 2 diabetes mellitus within the year before screening (e.g., multiple hospitalizations related to diabetes mellitus and/or severe hypoglycemia for which the subject required 3rd party assistance).
5. Any severe, delayed sequela of diabetes mellitus, e.g., worsening end-stage renal disease, advanced coronary artery disease, or myocardial infarction within the year before screening, or autonomic peristaltic problems, e.g., gastroparesis.
6. Anticipated change in insulin used during the study (change in dosage is allowed, but change in type or brand of insulin will result in the subject being withdrawn from the study).
7. Inadequately controlled thyroid disease, defined as a TSH or free T4 value > the upper limit of normal.
8. BMI > 45 kg/m2.
9. Any clinically significant (in the opinion of the Investigator) hematology or chemistry test results at screening, including any liver function test > 3x the upper limit of normal (subjects with elevated bilirubin due to Gilbert syndrome are eligible to participate).
10. Documented history of anti-insulin antibodies.
11. Treatment with glucocorticosteroids, immunosuppressants, or cytostatic agents within 60 days before screening (newly-prescribed or high-dose corticosteroids are prohibited; chronically administered oral, inhaled, topical, or intra-articular corticosteroids at a stable dosage are allowed if no increase in dose is anticipated during the study; See Appendix 3 [Section 17.3] for a list of allowed and prohibited concomitant medications).
12. Current use of medication intended to cause weight loss or weight gain.
13. Alcohol or substance use disorder within the 2 years before screening.
14. Any previous or anticipated treatment with interferons.
15. Any history of malignant disease within 5 years before screening, except for adequately treated basal cell carcinoma.
16. Severe concomitant physical or psychiatric diseases or conditions.
17. A history of a positive test result for HIV, hepatitis B, or hepatitis C; any subject who has a positive test result during the study may continue at the discretion of the Investigator.
18. Any history of pancreatitis or pancreatectomy.
19. Any diagnosis or condition that requires the subject to undergo procedures that could decrease antibodies in plasma or that would require treatment with immunosuppressant agents.
20. Any condition e.g., splenectomy, autoimmune disease, or rheumatologic disease, that could affect immunologic responses, could indicate an altered immune system, or could require treatment with a prohibited medication.
21. Any unresolved infection or a history of active infection within 30 days before screening other than mild or viral illness (as judged by the Investigator).
22. Any other disease or condition that in the opinion of the Investigator could confound the study results or limit the subject's ability to participate in the study or comply with follow-up procedures; or any other factor that would indicate a significant risk of loss to follow up.
23. Intolerance or history of hypersensitivity to insulin glargine or any excipient of IP.
24. Inability or unwillingness to wear the CGM sensor as required for the study, or to comply with the concomitant medication requirements in the FreeStyle Libre Pro Indications and Important Safety Information, during the CGM periods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Lu, PhD, Study Director — Gan & Lee Pharmaceuticals, USA; Elena A. Christofides, MD, FACE, Principal Investigator — Endocrinology Research Associates, Inc.
Locations (57):
- United States (57):
  - Simon Williamson Clinic, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Terence T. Hart, MD, Tuscumbia, Alabama
  - Family Practice Specialists, Phoenix, Arizona
  - Valley Research, Fresno, California
  - The Rose Salter Medical Research Foundation, Newport Coast, California
  - California Medical Research Association, Northridge, California
  - Northern California Research Corp., Sacramento, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Meridien Research, Bradenton, Florida
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Homestead Associates in Research, Homestead, Florida
  - Biotech Pharmaceutical Group, LLC, Miami, Florida
  - Genoma Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Peninsula Research, Ormond Beach, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Sestron Clinical Research, Marietta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Cedar Crosse Research Center, Chicago, Illinois
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - ActivMed Practices and Research - Methuen, Methuen, Massachusetts
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Physicians East, PA, Greenville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Endocrinology Associates, Inc., Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Mountain View Clinical Research, Greer, South Carolina
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - ClinSearch - Clinical Research Specialists, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Texas Diabetes & Endocrinology - Central Austin, Austin, Texas
  - Texas Diabetes & Endocrinology - South Austin, Austin, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Texas Diabetes & Endocrinology - Round Rock, Round Rock, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, Schertz, Texas
  - Radiant Research, Murray, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Stonesifer Clinical Research, Federal Way, Washington
  - Rainier Clinical Research Center, Inc., Renton, Washington
  - Clinical Investigations Specialists-Wisconsin, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Reviewed and approved by each IRB.
Pre-assignment Details: Inclusion and Exclusion Criteria.
Period: Safety Analysis Set
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Started | 284 | 283
Completed | 281 | 282
Not Completed | 3 | 1
Period: Completers
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Started | 281 | 282
Completed | 259 | 256
Not Completed | 22 | 26

BASELINE CHARACTERISTICS:
Population: All Subjects Assigned randomly to treatment (full analysis set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus® | Total
Number analyzed (Participants) | 284 | 283 | 567
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 163 | 178 | 341
  >=65 years | 121 | 105 | 226
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 122 | 226
  Male | 180 | 161 | 341
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 69 | 128
  Not Hispanic or Latino | 223 | 213 | 436
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 15 | 12 | 27
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 35 | 36 | 71
  White | 227 | 225 | 452
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: Participants]
  United States | 284 | 283 | 567
AIA result [Count of Participants; unit: Participants] — Presence or Absence of Confirmed, Positive, Anti-Insulin Antibody (AIA).
  Participants
    Negative | 252 | 263 | 515
    Positive | 5 | 1 | 6
    Nonreportable | 27 | 19 | 46
Body Mass Index (BMI) ≤45 kg/m^2 [Mean (Standard Deviation); unit: kg/m2] | 33.49 (5.589) | 33.59 (6.025) | 33.54 (5.806)
Duration of Diabetes (Years) [Mean (Standard Deviation); unit: Years] | 15.2 (7.96) | 15.3 (7.92) | 15.3 (7.93)
HbA1c (%) [Mean (Standard Deviation); unit: HbA1c (%)] — The baseline measure values of Glycosylated hemoglobin (HbA1c).
  HbA1c (%) | 8.49 (1.027) | 8.51 (1.029) | 8.50 (1.027)
NAb result [Count of Participants; unit: Participants] — Neutralizing antibody was tested only if the AIA result was positive. Subjects whose AIA result was negative or whose sample was defrosted or had temperature excursion were not tested for NAb.
  Participants
    Negative | 5 | 1 | 6
    Positive | 0 | 0 | 0
    Not Tested | 279 | 282 | 561
Thyroid Disease [Count of Participants; unit: Participants]
  Absence | 243 | 229 | 472
  Presence | 41 | 54 | 95
  Hypothyroidism | 34 | 45 | 79
  Hyperthyroidism | 2 | 0 | 2
  Structural abnormality | 1 | 1 | 2
  Thyroid Cancer | 0 | 0 | 0
  Other | 4 | 8 | 12
Weight (kg) [Mean (Standard Deviation); unit: Weight (kg)] | 98.011 (20.0532) | 98.141 (20.5269) | 98.076 (20.2732)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-induced Anti-Insulin Antibody (TI-AIA) is the Primary Endpoint
Description: Subjects were classified as experiencing a TI-AIA or not. A TI-AIA is defined as a subject experiencing a newly confirmed positive AIA status, if they were negative at baseline or a 4-fold increase in their titer values if they were positive. The primary outcome measure is summarized as the percent of subjects experiencing a TI-AIA in the group.
Time Frame: Baseline to Week 26
Population: The Safety Analysis Set (SS) was comprised of all subjects whose treatment assignment was randomly assigned who received any of the study treatment, even a partial dose, and had non-missing values.
Measure: Number; unit: Percentage of subjects with TI-AIA
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 281 | 282
Percentage of subjects with TI-AIA | 54 | 60
Statistical Analysis 1: Comparison: Gan & Lee Insulin Glargine Injection vs Lantus®; This is a two-arm study; Test type: Equivalence — The determination of equivalence was defined by the US-FDA as a confidence interval that was contained within the equivalence limits of +/- 10.7; Risk Difference (RD) = -2.1, 90% CI 2-sided [-7.6 to 3.5], Standard Error of Mean 3.39 — The asymptotic standard error was planned and is reported above

2. Secondary Outcome: CFB in HbA1c to Week 26
Description: Change is HbA1c value at week 26 minus the value at baseline.
Time Frame: Baseline to Week 26
Population: The Full Analysis Set (FAS) was comprised of all subjects whose treatment assignment was randomly assigned with non-missing baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 284 | 283
Percentage of glycosylated hemoglobin | -0.39 (0.079) | -0.45 (0.079)

3. Secondary Outcome: Immunogenicity - Percentage of Subjects in Each Treatment Group With Negative AIA at Baseline Who Develop Confirmed Positive AIA After Baseline
Description: The percentage of subjects in each treatment group with negative AIA at baseline who develop confirmed positive AIA after baseline and up to visit Week 26.
Time Frame: Baseline to Week 26
Population: Subset of subjects whose baseline AIA was negative (n=511).
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 249 | 262
Participants | 42 | 53

4. Secondary Outcome: Immunogenicity - Percentage of Subjects in Each Treatment Group With Confirmed Positive AIA at Baseline Who Developed at Least a 4-fold Increase in Titers After Baseline
Description: The percentage of subjects in each treatment group with confirmed positive AIA at baseline (n=6) who developed an important increase (at least a 4-fold increase in titers after baseline) up to visit Week 26.
Time Frame: Baseline to Week 26
Population: Subset of subjects in each treatment group with confirmed positive AIA at baseline (n=6).
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 5 | 1
Participants | 0 | 0

5. Secondary Outcome: Immunogenicity - Mean Change From Baseline in Each Treatment Group in AIA Titers After Baseline
Description: The mean change from baseline in each treatment group in AIA titers after baseline and up to visit Week 26.
Time Frame: Baseline to Week 26
Population: Subjects with Confirmed Positive Anti-Insulin Antibodies at Baseline with non-missing post-baseline AIA titer values (n=3).
Measure: Mean (Standard Deviation); unit: Titers
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 2 | 1
Titers | 23.5 (19.09) | -3.0 (NA) — The calculation of standard deviation for a subset of subjects of size 1 is undefined and therefore reporting standard deviation is not applicable.

6. Secondary Outcome: Immunogenicity - Percentage of Subjects With Confirmed Positive AIA After Baseline Who Develop Any Anti-insulin Neutralizing Antibodies After Baseline
Description: The percentage of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26 who develop any anti-insulin neutralizing antibodies after baseline and up to visit Week 26.
Time Frame: Baseline to Week 26
Population: Percentage of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26.
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 10 | 16
Participants | 1 | 3

7. Secondary Outcome: Immunogenicity - Percentage of Subjects With Confirmed Positive AIA After Baseline
Description: The percentage of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26.
Time Frame: Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 281 | 282
Participants | 58 | 61

8. Secondary Outcome: Efficacy - Postbaseline FBG Control
Description: The number and percentage of subjects who achieve an FBG test result of ≤ 8.0 mmol/L (≤ 144.0 mg/dL) at visit Week 26.
Time Frame: Baseline to Week 26
Population: FBG control (FBG ≤ 8.0 mmol/L)
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 284 | 283
Participants
  Lack of Postbaseline FBG control | 151 | 145
  Sufficient Postbaseline FBG control | 133 | 138

9. Secondary Outcome: Efficacy - HbA1c Control
Description: The number and percentage of subjects who achieve a HbA1c of < 7.0% at visit Week 26.
Time Frame: At Week 26
Population: HbA1c control (HbA1c < 7.0%)
Measure: Count of Participants; unit: Participants
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
Number analyzed (Participants) | 284 | 283
Participants
  Lack of Postbaseline HbA1c Control | 249 | 246
  Sufficient Postbaseline HbA1c Control | 35 | 37

ADVERSE EVENTS:
Time Frame: 26-weeks
Description: All untoward events, All-Cause Mortality, Serious, or Any Other (non-serious) Adverse Events were collected by regular investigator assessment and participants self-report, monitored, assessed, coded, and summarized.
Arm/Group | Gan & Lee Insulin Glargine Injection | Lantus®
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/282
Serious Adverse Events (participants affected / at risk) | 15/281 | 16/282
Other Adverse Events (participants affected / at risk) | 125/281 | 122/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gan & Lee Insulin Glargine Injection (N=281) | Lantus® (N=282)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Angina pectoris (General disorders) | 0 (0) | 1 (1)
Angina unstable (General disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
B-cell small lymphocytic lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back pain (General disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertensive emergency (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lactic acidosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localised infection (General disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Endocrine disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Endocrine disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal cell carcinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gan & Lee Insulin Glargine Injection (N=281) | Lantus® (N=282)
Hypoglycemia (Metabolism and nutrition disorders) | 120 (831) | 117 (761)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Nervous system disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1)
Injection related (General disorders) | 1 (1) | 0 (0)
Other (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT03371108/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03371108/SAP_001.pdf
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03371108/ICF_002.pdf